CLINICAL TRIAL: NCT01784510
Title: Two or Six cm From Pylorus at Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel-Raouf El-Geidie, assistant professor of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 3696
Record Dates: First submitted 2013-02-02; First posted 2013-02-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 2 cm (Active Comparator)
  Interventions: Procedure: distance of dissection of gastrocolic ligament from pylorus
- 6 cm (Experimental)
  Interventions: Procedure: distance of dissection of gastrocolic ligament from pylorus

INTERVENTIONS:
Procedure: distance of dissection of gastrocolic ligament from pylorus

SUMMARY:
Randomized controlled trial comparing between two technique of laparoscopic sleeve gastrectomy for treatment of morbid obesity. In the first technique the investigators started dissection of gastrocolic ligament 6 cm from pylorus and in the second one the distance was only 2 cm. The main primary outcome measure was weight loss.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity with body mass index more than 40 or 35 with at least one comorbidity

Exclusion Criteria:

* extreme of age less than 18 or over 65 years contraindications to laparoscopy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 months postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Surgical Center, Al Mansurah, Dakahlia Governorate, Egypt